CLINICAL TRIAL: NCT05080660
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY3526318 for the Treatment of Osteoarthritis Pain
Brief Title: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17592; H0P-MC-OA02 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-10-10; First posted 2021-10-18 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3526318 (Experimental): Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
  Interventions: Drug: LY3526318
- Placebo (Placebo Comparator): Participants received placebo orally, once daily, for 8-weeks treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally.
  Arms: LY3526318
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test safety and efficacy of study drug LY3526318 in for the treatment of knee pain due to with osteoarthritis (OA). This trial is part of the chronic pain master protocol H0P-MC-CPMP (NCT05986292) which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions for the duration of the study.
* Have presence of index knee pain for >12 weeks at screening.
* Have an x-ray supporting diagnosis of osteoarthritis according to the American College of Rheumatology with a Kellgren-Lawrence grade 2 to 4 radiographic classification of index knee.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have fibromyalgia
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Are in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Are largely or wholly incapacitated and unable to participate fully in all protocol procedures, for example, bedridden or confined to a wheelchair, permitting little or no selfcare.
* Have presence of surgical hardware or other foreign body in the index knee.
* Have an unstable index joint (such as a torn anterior cruciate ligament).
* Have had a surgical procedure or therapeutic injection in the affected knee within 3 months prior to starting the washout period.
* Have chronic pain syndrome, or other concurrent medical or arthritic conditions that could interfere with the evaluation of the index knee.
* Have a history of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, or amyloidosis.
* Have clinical signs and symptoms of active knee infection or crystal disease of the index knee.
* Have a history of infection in the index joint.
* Have a history of arthritis due to crystals (e.g., gout, pseudo gout).
* Have pain or functional impairment due to ipsilateral hip osteoarthritis.
* Are pregnant or breastfeeding.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (30):
- United States (28):
  - Synexus- Chandler, Chandler, Arizona
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Alliance for Multispecialty Research, LLC Tempe, Tempe, Arizona
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - Synexus Clinical Research US, Inc - Orlando, The Villages, Florida
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Synexus - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Synexus - US, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Chronic Pain Master Protocol (CPMP): A Study of LY3526318 in Participants With Osteoarthritis — https://trials.lillytrialguide.com/en-US/trial/o5FS87tuIKFcTChW9I2GN

RESULTS

PARTICIPANT FLOW:
Groups:
- 250 Milligram (mg) LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
Period: Overall Study
Arm/Group | 250 Milligram (mg) LY3526318 | Placebo
Started | 107 | 53
Received at Least One Dose of Study Drug (Safety Population Week 1-4) | 107 | 53
Safety Population Week 5-8 (All participants who took at least 1 dose of study drug and who did not discontinue at or prior to week 4.) | 99 | 51
Completed | 94 | 51
Not Completed | 13 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Non-compliance With Study Drug and Procedures | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Deviation | 2 | 0
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled or randomized participants who received at least one dose of study drug.
Groups:
- 250 mg LY3526318: Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks and were switched to placebo once daily for the next 4 weeks of the treatment period.
- Total: Total of all reporting groups
Arm/Group | 250 mg LY3526318 | Placebo | Total
Number analyzed (Participants) | 107 | 53 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 31 | 85
  >=65 years | 53 | 22 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.3) | 62.7 (9.3) | 63.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 33 | 101
  Male | 39 | 20 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 12 | 42
  Not Hispanic or Latino | 77 | 40 | 117
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 88 | 38 | 126
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 107 | 53 | 160
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine. Population: Participants with non-missing baseline NRS data.
  score on a scale
    number analyzed (Participants) | 106 | 53 | 159
    (all) | 5.52 (1.60) | 5.91 (1.25) | 5.65 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Posterior mean change from baseline, 95 percent (%) credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes number of participants with non-missing values at Week 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 97 | 52
score on a scale | -0.95 [-1.24 to -0.67] | -1.18 [-1.58 to -0.78]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.23, 95% CI 2-sided [-0.26 to 0.73] — Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes number of participants with non-missing values at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 51
score on a scale | -1.26 [-1.60 to -0.93] | -1.45 [-1.92 to -0.99]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.19, 95% CI 2-sided [-0.39 to 0.76] — Posterior mean difference with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline on the Western Ontario and McMaster University Arthritis Index (WOMAC®) Pain Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 5 questions on the pain subscale, and participants used a 0 to 4 Likert scale to answer each question for the current day: 0 = no pain, and 4 = extreme pain. The scores for the pain subscale were calculated by summing the scores of the questions for each participant at each time point. The range of possible scores is 0 to 20 for the pain subscale. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 107 | 52
score on a scale | -1.87 [-2.40 to -1.36] | -2.50 [-3.21 to -1.79]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.62, 95% CI 2-sided [-0.23 to 1.47] — Posterior mean difference with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline on the Western Ontario and McMaster University Arthritis Index (WOMAC®) Pain Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 5 questions on the pain subscale, and participants used a 0 to 4 Likert scale to answer each question for the current day: 0=no pain, and 4=extreme pain. The scores for the pain subscale were calculated by summing the scores of the questions for each participant at each time point. The range of possible scores is 0 to 20 for the pain subscale. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 51
score on a scale | -2.51 [-3.15 to -1.87] | -2.85 [-3.69 to -1.99]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.34, 95% CI 2-sided [-0.67 to 1.34] — Posterior mean difference with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline on the WOMAC® Stiffness Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 2 questions in the stiffness subscale and participants used a 0 to 4 Likert scale to answer each question for the current day: 0=no stiffness, and 4=extreme stiffness. The scores for each subscale were calculated by summing the scores of the questions in each respective subscale for each participant at each time point. The range of possible scores is 0 to 8 for the stiffness subscale.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 100 | 52
score on a scale | -1.04 [-1.32 to -0.76] | -1.11 [-1.48 to -0.75]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.08, 95% CI 2-sided [-0.35 to 0.50] — Posterior mean difference with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline on the WOMAC® Stiffness Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 2 questions in the stiffness subscale and participants used a 0 to 4 Likert scale to answer each question for the current day: 0 = no stiffness, and 4 = extreme stiffness. The scores for each subscale were calculated by summing the scores of the questions in each respective subscale for each participant at each time point. The range of possible scores is 0 to 8 for the stiffness subscale.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 51
score on a scale | -1.16 [-1.46 to -0.86] | -1.26 [-1.65 to -0.87]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.10, 95% CI 2-sided [-0.35 to 0.55] — Posterior mean difference with 95% credible interval is reported

7. Secondary Outcome: Change From Baseline on the WOMAC® Physical Function Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 17 questions in the physical function subscale, and participants used a 0 to 4 Likert scale to answer each question for the current day: 0=no difficulty, and 4=extreme difficulty. The scores for each subscale were calculated by summing the scores of the questions in each respective subscale for each participant at each time point. The range of possible scores is 0 to 68 for the physical function subscale.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 99 | 51
score on a scale | -6.48 [-8.21 to -4.76] | -8.46 [-10.86 to -6.10]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 1.98, 95% CI 2-sided [-0.88 to 4.88] — Posterior mean difference with 95% credible interval is reported

8. Secondary Outcome: Change From Baseline on the WOMAC® Physical Function Subscale
Description: as for outcome 7
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 95 | 50
score on a scale | -8.04 [-10.07 to -6.01] | -11.09 [-13.82 to -8.33]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 3.05, 95% CI 2-sided [-0.29 to 6.38] — Posterior mean difference with 95% credible interval is reported

9. Secondary Outcome: Change From Baseline in Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1=very much better, and 7=very much worse.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 100 | 52
score on a scale | 3.18 [2.97 to 3.40] | 3.05 [2.75 to 3.35]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.13, 95% CI 2-sided [-0.23 to 0.50] — Posterior mean difference with 95% credible interval is reported

10. Secondary Outcome: Change From Baseline in Overall Improvement as Measured by Patient's Global Impression of Change
Description: as for outcome 9
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 51
score on a scale | 2.96 [2.74 to 3.18] | 2.97 [2.66 to 3.28]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.01, 95% CI 2-sided [-0.39 to 0.37] — Posterior mean difference with 95% credible interval is reported

11. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used during the preliminary data entry period and daily throughout the study to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 97 | 52
score on a scale | -1.08 [-1.38 to -0.79] | -1.38 [-1.79 to -0.97]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.30, 95% CI 2-sided [-0.21 to 0.81] — Posterior mean difference with 95% credible interval is reported

12. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 51
score on a scale | -1.41 [-1.76 to -1.05] | -1.70 [-2.19 to -1.21]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.29, 95% CI 2-sided [-0.31 to 0.90] — Posterior mean difference with 95% credible interval is reported

13. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0=no pain, and 100=worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 100 | 52
score on a scale | -11.69 [-15.47 to -7.87] | -17.82 [-23.08 to -12.61]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 6.14, 95% CI 2-sided [-0.24 to 12.52] — Posterior mean difference with 95% credible interval is reported

14. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: as for outcome 13
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 51
score on a scale | -16.41 [-20.55 to -12.32] | -21.55 [-27.30 to -15.81]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 5.15, 95% CI 2-sided [-1.90 to 12.18] — Posterior mean difference with 95% credible interval is reported

15. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Question 1 asks time to fall asleep and it is reported in 5-point timeframe categories. Question 2 asks average hours of sleep. In the remaining 10 questions participants report how often a sleep symptom or problem was present on a scale ranging from '0=all of the time' to '5=none of the time.' MOS Sleep scale dimension scores range from 0 to 100 with lower score indicating improvement, except for the dimension of sleep adequacy, where higher scores indicate improvement. Here, the average hours of sleep (i.e., Question 2) is reported as the average number of hours slept each night during the past week (range 0 to 24 hours). Higher number of hours slept indicates improvement.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 100 | 52
Hours per night | 0.04 [-0.14 to 0.22] | 0.06 [-0.18 to 0.31]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.02, 95% CI 2-sided [-0.32 to 0.27] — Posterior mean difference with 95% credible interval is reported

16. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: as for outcome 15
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Hours per night
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 50
Hours per night | -0.01 [-0.21 to 0.19] | 0.19 [-0.08 to 0.45]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.20, 95% CI 2-sided [-0.52 to 0.13] — Posterior mean difference with 95% credible interval is reported

17. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: Total amount of rescue medication use as measured by average daily dosage. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mg per day (mg/day)
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 97 | 52
mg per day (mg/day) | 271.27 [182.84 to 359.36] | 172.92 [47.39 to 296.22]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 98.35, 95% CI 2-sided [-51.95 to 250.88] — Posterior mean difference with 95% credible interval is reported

18. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: as for outcome 17
Time Frame: Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: mg/day
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 90 | 51
mg/day | 284.83 [185.06 to 385.02] | 161.47 [22.36 to 299.42]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = 123.36, 95% CI 2-sided [-46.51 to 293.69] — Posterior mean difference with 95% credible interval is reported

19. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) (United States)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health: 0=a health state equivalent to death, and 1=perfect health.
  Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 4
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 100 | 52
score on a scale | 0.04 [0.00 to 0.08] | 0.05 [-0.01 to 0.10]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.01, 95% CI 2-sided [-0.06 to 0.05] — Posterior mean difference with 95% credible interval is reported

20. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) (United States)
Description: as for outcome 19
Time Frame: Baseline, Week 8
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 250 mg LY3526318 | Placebo
Number analyzed (Participants) | 96 | 51
score on a scale | 0.05 [0.00 to 0.10] | 0.05 [-0.01 to 0.12]
Statistical Analysis 1: Comparison: 250 mg LY3526318 vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.00, 95% CI 2-sided [-0.07 to 0.07] — Posterior mean difference with 95% credible interval is reported

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: All participants under the safety population for week 1-4 and week 5-8.
Groups:
- 250 mg LY3526318 (Week 1 to 4): Participants received 250 mg of LY3526318 orally, once daily for the first 4 weeks of treatment period (Week 1-4).
- 250 mg LY3526318/Placebo (Week 5 to 8): Participants who received 250 mg of LY3526318 in the first 4 weeks were switched to received placebo once daily for the next 4 weeks of the treatment period (Week 5-8).
- Placebo (Week 1 to 4): Participants received placebo orally, once daily, for week 1 to 4 of treatment period.
- Placebo (Week 5 to 8): Participants received placebo orally, once daily, for week 5 to 8 of treatment period.
Arm/Group | 250 mg LY3526318 (Week 1 to 4) | 250 mg LY3526318/Placebo (Week 5 to 8) | Placebo (Week 1 to 4) | Placebo (Week 5 to 8)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/99 | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/107 | 0/99 | 1/53 | 0/51
Other Adverse Events (participants affected / at risk) | 31/107 | 13/99 | 21/53 | 8/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg LY3526318 (Week 1 to 4) (N=107) | 250 mg LY3526318/Placebo (Week 5 to 8) (N=99) | Placebo (Week 1 to 4) (N=53) | Placebo (Week 5 to 8) (N=51)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 250 mg LY3526318 (Week 1 to 4) (N=107) | 250 mg LY3526318/Placebo (Week 5 to 8) (N=99) | Placebo (Week 1 to 4) (N=53) | Placebo (Week 5 to 8) (N=51)
Headache (Nervous system disorders) | 6 | 1 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Persistent genital arousal disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Anti-muscle specific kinase antibody (Investigations) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Hepatitis B surface antibody positive (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Uterine leiomyoma*a (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Allergy to metals (Immune system disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT05080660/Prot_004.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT05080660/SAP_005.pdf